CLINICAL TRIAL: NCT04310683
Title: The Live Birth Rate in Natural Cycle or Stimulated Cycle Versus Hormone Replaced Cycle in Patients Undergoing Frozen-thawed Embryo Transfer
Brief Title: Natural Cycle or Stimulated Cycle Versus Hormone Replaced Cycle for Pre-eclampsia Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREECLAMPSIA
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural cycle for endometrium preparation (Other): patients will have ovulation before embryo transfer
  Interventions: Other: natural cycle for endometrium preparation
- hormone replaced cycle for endometrium preparation (Experimental): patients will do not have ovulation before embryo transfer
  Interventions: Other: hormone replaced cycle for endometrium preparation

INTERVENTIONS:
Other: natural cycle for endometrium preparation — patients will not use oral contraceptive drugs
  Other Names: non
  Arms: natural cycle for endometrium preparation
Other: hormone replaced cycle for endometrium preparation — patients will receive oral contraceptive drugs for menstruation before embryo transfer
  Other Names: non
  Arms: hormone replaced cycle for endometrium preparation

SUMMARY:
Recent sutdies indicate that the existence of corpus lutein in the ovary is a key point to prevent preeclampsia, and patients undergoing FET with hormone replaced cycle have no corpus lutein and the absence of corpus lutein significantly increases the risk of preeclampsia in these patients. We aim to conduct a single center randomized trial study to compare the preeclampsia rate between the natural cycle and the hormone replaced cycle in patients undergoing FET.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 42 years old women;
2. normal ovulation;
3. Scheduled to undergo frozen-thawed embryo transfer.
4. Agreeing with the informed consent.

Exclusion Criteria:

1. Those who experienced embryo transfer cycle failure for at least three times;
2. One or both of the ovaries removed;
3. Hypertention disease before embryo transfer;
4. No available embryo for transfer
5. Oocyte or sperm donated cycles

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 840 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
live birth rate | delivery
  A delivery is considered successful live birth

SECONDARY OUTCOMES:
pre-eclampsia | From gestational week 20 to delivery
  Preeclampsia is defined using the current American College of Obstetricians and Gynecologists definitions (Gynecologists; and Pregnancy 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhang, M.D. Ph.D., Principal Investigator — Women's Hospital School Of Medicine Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided